CLINICAL TRIAL: NCT06620692
Title: A Phase IIa Study to Investigate the Efficacy and Safety Profile of GM-XANTHO [GM-XAN003] in Patients with Psoriasis
Brief Title: A Study to Investigate the Efficacy and Safety Profile of GM-XANTHO [GM-XAN003] in Patients with Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xantho Biotechnology Co., LTD (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XANGMXH20211027
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 % GM-XANTHO [GM-XAN003] group (Experimental): Patients will take the test product, 5 % GM-XANTHO [GM-XAN003].
  Interventions: Drug: 5% GM-XANTHO [GM-XAN003]
- Placebo group (Placebo Comparator): Patients will take the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5% GM-XANTHO [GM-XAN003] — 5% GM-XANTHO [GM-XAN003]
  Arms: 5 % GM-XANTHO [GM-XAN003] group
Drug: Placebo — The placebo
  Arms: Placebo group

SUMMARY:
This trial is a Phase IIa clinical trial. Around 65 subjects will be enrolled into this study to primarily assess the treatment efficacy of 5% GM-XANTHO in patients with psoriasis, as well as the safety and tolerability of 5% GM-XANTHO. Two third of the total subjects will be given the investigational product, 5% GM-XANTHO, and the other third will take placebo. The treatment period will last for 28 consecutive days, followed by a safety follow-up for 2 weeks. During the study, there will be 8 scheduled visits to the clinical center.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients are ≥ 20 years old.
2. Patients who are able to understand the nature of this study and accept to enter the study by signing written informed consent.
3. Patients are willing or able to comply with procedures required in this protocol including self-administration of study drug.
4. Patients who have well diagnosed chronic plaque psoriasis for at least 6 months before the Screening Visit (according to Am Fam Physician. 2013 May 1;87(9):626-633).
5. The severity of plaque psoriasis is stable mild to moderate which meets the following disease activity criteria at both Screening and Baseline Visit (according to Joint AAD-NPF Guidelines)
6. Patients who agree discontinuation of systemic corticosteroids and systemic immune modulating agents during the study period.
7. Patients who agree discontinuation of all local treatment modalities, including but not limited to topical corticosteroid or light treatments during the study period for/on the affected regions.
8. Patients are required to stop using treatment modalities listed in Criteria #6 and #7 at least 14 days (or longer if the treatment half-life requires so; 7 half-life should have elapsed).
9. Patients have adequate hematopoietic, hepatic function, and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin ≥ 10 g/dL
   * Total WBC ≥ 3,000 cells/μL
   * Platelet ≥ 55,000 counts/μL without transfusion support
   * Total bilirubin ≤ 1.5× ULN and no sign of jaundice
   * ALT and AST ≤ 5× ULN and no clinical significance
   * Creatinine ≤ 1.5× ULN and no clinical significance
10. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods shown below, for during and at least 4 weeks after GM-XANTHO [GM-XAN003] treatment.

    1. Total abstinence [when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
    2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male sterilization. For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
    4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

    d.1 Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

    d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

1. Patients with the following subtype of psoriasis:

   * Erythrodermic psoriasis
   * Generalized or localized pustular psoriasis,
   * edication-induced or medication-exacerbated psoriasis,
   * New onset guttate psoriasis.
2. Patients who have any concurrent skin condition that will interfere with assessment of treatment.
3. Patients who have systemic infection during the last 2 weeks prior to Screening Visit or active infection on the psoriasis lesion.
4. Patients who have known hypersensitivity to the study medication.
5. Patients with chronic condition(s) which either is not stable or not well controlled.
6. Patients having positive results for HBV, HCV or HIV screens.
7. Patients who are pregnant or breast feeding.
8. Patients who have the medical history of malignancy of any organ system (other than cervical carcinoma in situ or successfully treated non-melanoma skin cancer) within 5 years prior to study entry.
9. Patients had participated in investigational drug trials and took any investigational drugs within 30 days or within 5 half-life of the investigational drugs prior to the screening visit.
10. Patients who are not suitable to participate in the trial as judged by the Investigator(s).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Psoriasis Area and Severity Index (PASI) | through study completion, an average of 7 weeks

SECONDARY OUTCOMES:
Change from baseline in Body Surface Area (BSA) affected | through study completion, an average of 7 weeks
Change from baseline in quality of life by using the Dermatology Life Quality Index (DLQI) | through study completion, an average of 7 weeks
Incidence of subjects experiencing treatment related AE with ≥ Grade 2 according to the predefined toxicity grading scale in this study | through study completion, up to 2 years
Number of patients achieving PGA of 0 or 1 at each visit | through study completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical PM, Study Director — Xantho Biotechnology Co., LTD

IPD SHARING:
Plan to Share IPD: No